CLINICAL TRIAL: NCT04145154
Title: Effect of the Rich Plasma in Growth Factors on the Cicatrization of Diabetic Ulcers
Brief Title: Plasma and Scarring of Diabetic Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, María Guadalupe de Lourdes González Avalos, Principal investigator, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Plasma
Record Dates: First submitted 2019-10-22; First posted 2019-10-30 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Chronic Skin Ulcer; Diabetic Foot; Plasma Protein; Transport Protein
Keywords: Platelet; Diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma (Experimental): Subjects to whom platelet rich plasma is applied
  Interventions: Other: Application of platelet rich plasma in chronic wounds of diabetic origin
- Advanced cure (No Intervention): Subjects to whom advanced healing is performed

INTERVENTIONS:
Other: Application of platelet rich plasma in chronic wounds of diabetic origin — Application of plasma rich in autologous growht factors after advanced healing
  Other Names: Advanced cure
  Arms: Plasma

SUMMARY:
Diabetic foot is defined by World Health Organization as a syndrome in which the presence of neuropathy, ischemia and infection cause tissue damage or ulcers from minor trauma. This condition can be controlled in its early stages with conservative treatment, which is effective in preventing infections and amputations. However, even with the new knowledge acquired and the development of new therapies, the specialist often faces wounds that do not improve despite the proper treatment, so therapies have been sought to help the healing of these Ulcers. Growing evidence suggests that healing of chronic diabetic foot ulcers depends on growth factors and that the therapeutic use of these in wounds has the potential to accelerate their healing in conjunction with wound care Conventional. This study evaluates the effect of plasma rich in autologous growth factors on healing chronic ulcers of diabetic origin.

This is a randomized clinical trial that evaluates two study groups. Control group in which advanced weekly healing will be performed while the post-advanced healing study group will be performed the intradermal application of plasma rich in growth factors. These manoeuvres will be performed once a week for four weeks and at the end of the study the results in both groups will be checked. Both groups will also evaluate, frequency and intensity of pain, quality of life, histological changes in ulcers and metabolic evaluation

DETAILED DESCRIPTION:
The diabetic foot is a devastating complication of diabetes mellitus that is accompanied by chest-evolving ulcers, which often lead to amputation. Annually more than a million people lose some limb stake because of this cause. Foot ulceration is the most common complication of diabetic patients and is thought to affect up to 15% of them throughout their lives (8, 9).

Ulcers that do not progress over a period of approximately 4 weeks should be reassessed. Several studies have also shown that chronic ulcers in general and diabetic foot ulcers in particular have alterations in fibroblast proliferation, the balance between growth factors, metalloproteinase (MMP) and remodeling extracellular matrix (2, 8, 9).

Changes in matrix metalloproteinase levels, as well as Regulated on Activation , Normal T-cell Expressed and Secretated, interleukin and procalcitonin have been correlated with wound healing (10). Metalloproteinase and its regulators, matrix metalloproteinase tissue inhibitors (TIMPes) are necessary for a wound to be properly healed at an appropriate level, at the right location and for a precise period of time. These aspects, it is presumed, are not met in chronic wounds such as ulcers of diabetic origin (11).

Autologous growth factor-rich plasma (PRFC), applied at the wound site releases dozens of growth factors, chemokines and cytokines that regulate angiogenesis, epithelialization and regeneration (15, 16). They are secreted by the granules and has been found to contribute to increase the speed of the natural healing process with a decrease in time (4).

Platelet-rich plasma is defined as an autologous or allogeneic platelet derivative with a concentration of platelets higher than the baseline. Autologous growth factor-rich plasma (PRFC) is the fraction of plasma derived from autologous blood, which after being processed by centrifugation, has a higher concentration of platelets and higher than baseline growth factors (8). There are two obtaining techniques: closed and open. In the case of obtaining by "closed technique", the method used must follow the instructions described in the disposable kits used in each commercial system. The "open technique" allows, on the other hand, from lower blood volumes and simple equipment, to obtain a higher concentration of growth factors (25).

Given its autologous nature, PRFC is a safe product, which by definition lacks the potential risk of disease transmission involving the use of donor blood material. With regard to the oncogenic potential of PRFC that some authors have suggested, there is no available evidence to support it.

Key factors released include platelet-derived growth factor (PDGF), beta transforming growth factor (TGF-b), platelet factor 4 (PF4), interleukin 1 (IL-1), the angiogenic factor derived from platelets (PDAF), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet-derived endothelial growth factor (PDEGF), epithelial cell growth factor (ECGF), insulin (IGF-1), osteocalcin, osteonectin, fibrinogen, fibronectin and thrombospondin (TSP) (11,27). These proteins secreted by activated platelets influence many aspects of healing.

PRFC has been used in different areas of Regenerative Medicine to improve wound healing processes with multiple clinical applications in different fields of medicine: General Surgery, Traumatology and Sports Medicine, Dentistry and Surgery Plastic and Reconstructive Surgery, Dermatology, Neurology and Neurosurgery (28, 8).

The implementation of new strategies in the treatment of diabetic foot ulcers involving growth factors and platelet-rich plasma (15,16,17,20,27,28) has a history of basing it.

Despite these solid biological bases, the treatment results of skin ulcers with platelet-derived growth factors are varied and there are relatively few controlled studies. There is confusion about the usefulness of platelet-rich plasma because the studies that have evaluated them use a wide range of products (different concentrations of platelets and leukocytes, different techniques and frequencies of application, different types of injuries to be treated, very heterogeneous and different endpoints) that make it almost impossible to compare data and draw conclusions (29, 30).

There are reviews that evaluate the results that have been had so far on the effects that these biological supplements with platelets offer as adjuvants in wound healing and healing. A meta-analysis published in 2016, which included 10 randomized clinical trials evaluating the effect of PRFC on chronic wound healing. Three of these randomized clinical trials involved ulcers of diabetic origin and three studies involved venous leg ulcers. The overall analysis did not shed light on the effectiveness of PRFC, but the results indicated that autologous PRFC can improve the healing of diabetic ulcers compared to standard care, although the value of evidence is low (46).

This is why we believe it is appropriate to carry out studies that allow to evaluate in a clear way and with a simple but complete description the effect that the use of PRFC has on the healing of chronic ulcers of diabetic origin of difficult management.

Research hypothesis. The 4-week intradermal application of Plasma rich in growth factors (PRFC) reduces healing time of chronic ulcers of difficult-to-manage diabetic origin, the size of the injury, induces changes at the level histological and contributes to reducing pain and improving the patient's quality of life compared to the best treatment available.

Material and methods. Randomized clinical trial conducted in patients with chronic ulcers (more than 4 weeks of evolution) of diabetic origin that come to the Wound Clinic of the Regional General Hospital of León for evaluation and care.

The sample size was calculated in 20 patients per group (control group and study group), to detect at least a 50% difference in the reduction in the dimensions of the chronic ulcer at the end of the manoeuvre, with a statistical significance of 0.05% and a poten 80%. Patients will be selected by non-probabilistic sampling for convenience.

Procedure. Patients will be incorporated into the study through the Wound Clinic and the Hematology department of the Regional General Hospital of León where they will be invited to participate in it, after explanation of the procedure and those who accept, they will be invited will request to sign informed consent. Patients who agree to participate in the study will have metabolic and haematological evaluation by the Hematology service of the same hospital. Laboratory studies (hematic biometrics, blood chemistry, HbA1C, lipid profile and coagulation times) will be performed. Patients will be cited 1 time per week at the Wound Clinic and advanced ulcer cure will be performed in both groups consisting of healing with physiological and antiseptic solution, biofilm debridement, as well as devitalized tissue, occluding with non-absorbent gauze, dried gauze and bandage in both groups. The study group will also have the intradermal application of PRFC after healing. The study group will also be taken as a biopsy by punch (5mm x 5mm, considering a small part) in the first week (before the application of PRFC) and at the end of treatment (1 week after the last application of prFC). In patients where a complete ulcer closure is achieved, no final biopsy taken to prevent further ulceration from occurring. This in order to determine the effects of Plasma rich in growth factors at the histological level on ulcers of diabetic origin. Such procedures shall be carried out by the student. During each appointment, prior to the completion of the treatment, the measurement of the ulcer in its major and smallest diameters will be performed and the area will be calculated through computerized planimetry. This will be done by the surgeon general and responsible for the Wound Clinic who will be blinded which group each patient belongs to). Each patient will also be evaluated through the Visual Pain Analog Scale (EVA) and the SF-12 Lifestyle Questionnaire, each week. Both scales with validity in force (49, 50). During the duration of the study, weekly photographic monitoring of ulcers will be carried out to assess their evolution and response to treatment in each patient. Both the evaluations and the photographic follow-up will be carried out by the student.

Technical of centrifugation and obtaining PRFC. After 8 hours fasting, blood sampling (20 cc) will be performed by ulnar artery puncture, which will be collected in sterile tubes with sodium citrate at 3.8% as anticoagulant. A sample will be used to perform a pre-centrifugation platelet count. The rest of the blood sample will be centrifuged at 3200 revolutions per minute (rpm) for 15 minutes at room temperature; separation by pipetting of the obtained plasma (approximately 3-4 ml) with a variable platelet content, which will be centrifuged again for 8 minutes at 1800 rpm, at room temperature. Subsequently by meticulous pipetting, the fractions obtained from the plasma shall be separated from above, and collected in sterile tubes separated in such a way that the last fraction obtained (approximately 1-5 to 2 ml and located in the lower portion of the tube) corresponding to the plasma rich in growth factors or PRFC (26). A 0.5 ml sample will be taken from this fraction of PRFC to perform a platelet count and determine post-centrifugation platelet performance in each patient and application. This value will be recorded to determine the increase in platelet concentration in each patient. The remaining fraction (1.5 ml) will be applied through intradermal injection immediately upon collection. This procedure will be performed in the Laboratory of the General Hospital of León by the same person trained and familiar with the procedure throughout the study. Calcium citrate will not be added as a activator as it is considered according to the literature that the activation of growth factors takes place in soft tissues once PRFC comes into contact with collagen fibers.

TECHNICAL APPLICATION OF PRFC Once the ulcer has been cured in the manner described above and before the application of the gauze, the study group will be applied to 2 thirds of the PRFC obtained through intradermal injection in tod or the perimeter of the ulcer with 3cc syringe and hypodermic needle. The remaining third will be applied to the ulcer bed by drip technique. Subsequently, non-absorbent gauze will be placed on it and finally covered with dried gauze and bandage. These will be removed until the next PRFC application (1 week).

Statistical Analysis. Continuous variables will be reported as means +/- standard deviations and categorical ones as frequencies and percentages. We will perform Student T for the initial comparison of the study groups and X2 according to the type of variable. To test our hypothesis we will perform ANOVA of repeated measurements and post hoc test of Tukey. A Multiple Correlation analysis will determine the possible association of other factors that influence the healing time of ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic ulcers of diabetic origin of more than 4 weeks of evolution in lower extremities with treatment with hypoglycemic and/or insulin.
* Age over 18 years and under 75 years, both genders.
* Platelet count greater than 100,000 platelets per mm3.
* Serum Hb level of > 9 g/dl both genders and<18 g/dl in men and <16 g/dl in women.
* HbA1c level <8%
* Serum triglyceride level <300 mg/dl.
* Grade IA and IIA ulcers according to Texas classification.
* Dimension greater than 3 cm in any of its diameters. 9. Ankle-arm index >0.7.

Exclusion Criteria:

* Chronic ulcers of traumatic, neoplastic, infectious, vascular and ischemic origin.
* Evidence of malignant ulcer
* Clinical evidence of ulcer infection at the start of treatment such as purulent secretion, local hyperthermia or active systemic infection.
* Haematological or coagulation disturbances.
* Carriers of syphilis, HIV, Hepatitis Virus B and C.
* Chronic use of corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Changing the dimensions of the ulcer area | Up to four weeks
  The area of the ulcers will be measured every week in both groups in square centimeters recording the change

SECONDARY OUTCOMES:
Change in the major and minor diameters of ulcers | Up to four weeks
  The largest and smaller diameters will be measured in centimeters each week in both groups
Change in pain intensity | Up to four weeks
  The change in pain intensity will be measured in both groups each week through.It is evaluated using the Pain Analogue Scale, where 0 is no pain and 10 is the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: GLORIA B SABANERO, DOCTOR, Study Director — Universidad de Guanajuato
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazaro-Martinez JL, Garcia-Morales E, Beneit-Montesinos JV, Martinez-de-Jesus FR, Aragon-Sanchez FJ. [Randomized comparative trial of a collagen/oxidized regenerated cellulose dressing in the treatment of neuropathic diabetic foot ulcers]. Cir Esp. 2007 Jul;82(1):27-31. doi: 10.1016/s0009-739x(07)71657-3. Spanish. PMID 17580028
- [Background] Piccin A, Di Pierro AM, Canzian L, Primerano M, Corvetta D, Negri G, Mazzoleni G, Gastl G, Steurer M, Gentilini I, Eisendle K, Fontanella F. Platelet gel: a new therapeutic tool with great potential. Blood Transfus. 2017 Jul;15(4):333-340. doi: 10.2450/2016.0038-16. Epub 2016 Jul 25. PMID 27483482
- [Background] Suthar M, Gupta S, Bukhari S, Ponemone V. Treatment of chronic non-healing ulcers using autologous platelet rich plasma: a case series. J Biomed Sci. 2017 Feb 27;24(1):16. doi: 10.1186/s12929-017-0324-1. PMID 28241824
- [Background] Suresh DH, Suryanarayan S, Sarvajnamurthy S, Puvvadi S. Treatment of a non-healing diabetic foot ulcer with platelet-rich plasma. J Cutan Aesthet Surg. 2014 Oct-Dec;7(4):229-31. doi: 10.4103/0974-2077.150786. PMID 25722604
- [Background] Hahm G, Glaser JJ, Elster EA. Biomarkers to predict wound healing: the future of complex war wound management. Plast Reconstr Surg. 2011 Jan;127 Suppl 1:21S-26S. doi: 10.1097/PRS.0b013e3181fbe291. PMID 21200268
- [Background] Lindley LE, Stojadinovic O, Pastar I, Tomic-Canic M. Biology and Biomarkers for Wound Healing. Plast Reconstr Surg. 2016 Sep;138(3 Suppl):18S-28S. doi: 10.1097/PRS.0000000000002682. PMID 27556760
- [Background] Cervelli V, De Angelis B, Lucarini L, Spallone D, Balzani A, Palla L, Gentile P, Cerulli P. Tissue regeneration in loss of substance on the lower limbs through use of platelet-rich plasma, stem cells from adipose tissue, and hyaluronic acid. Adv Skin Wound Care. 2010 Jun;23(6):262-72. doi: 10.1097/01.ASW.0000363551.82058.36. PMID 20489388
- [Background] Singh B, Goldberg LJ. Autologous Platelet-Rich Plasma for the Treatment of Pattern Hair Loss. Am J Clin Dermatol. 2016 Aug;17(4):359-67. doi: 10.1007/s40257-016-0196-2. PMID 27234711
- [Background] Cobos R, Aizpuru F, Parraza N, Anitua E, Orive G. Effectiveness and efficiency of platelet rich plasma in the treatment of diabetic ulcers. Curr Pharm Biotechnol. 2015;16(7):630-4. doi: 10.2174/138920101607150427111926. PMID 25934972
- [Background] Savelyeva EN, Kudryavtsev AM. [AFLP Analysis of Genetic Diversity in the Genus Mallus Mill. (Apple)]. Genetika. 2015 Oct;51(10):1126-33. Russian. PMID 27169227
- [Background] Martinez-Zapata MJ, Marti-Carvajal AJ, Sola I, Exposito JA, Bolibar I, Rodriguez L, Garcia J, Zaror C. Autologous platelet-rich plasma for treating chronic wounds. Cochrane Database Syst Rev. 2016 May 25;2016(5):CD006899. doi: 10.1002/14651858.CD006899.pub3. PMID 27223580